CLINICAL TRIAL: NCT00188227
Title: Comparison of Three Different Pain and Anxiety Reducing Methods in Adult Patients Undergoing Bone Marrow Puncture
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CGC05MK1001
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2007-04-20 (Estimated); Status verified 2005-09

CONDITIONS: Patients Undergoing Puncture of the Bone Marrow
Keywords: Bone marrow puncture; Pain
MeSH Terms: conditions — Pain | interventions — Midazolam; Hypnotics and Sedatives; Pirinitramide

INTERVENTIONS:
Drug: Midazolam (sedative)
Drug: Piritramid (analgetic)
Behavioral: Cognitive exercises

SUMMARY:
The purpose of this study is to investigate and compare the effects of three different methods for reducing pain and anxiety in adult patients undergoing puncture of the bone marrow. The investigated methods are: cognitive behavioural technique, administration of a sedative drug(Midazolam) and administration of an analgetic drug (Piritramid)prior to the procedure. Additionally, there are two comparison groups in which the patients receive either placebo treatment or no treatment at all.

DETAILED DESCRIPTION:
The puncture of the bone marrow is a routine medical procedure which is often performed in the field of hematology/oncology. When carefully and appropriately performed, the puncture of the bone marrow has a very low rate of complications and is generally safe for the patient. However, it is an invasive and painful procedure associated with anxiety, especially in patients undergoing repeated punctures. Therefore an appropriate preparation of the patient for the puncture is essential in order to minimize the stress experienced during the procedure. In this regard, there are numbers of both pharmacological and non-pharmacological interventions in pedriatric patients aimed at reducing the punction related pain and anxiety in this patients. Nevertheless an evidence based approach for the pretreatment of the patients is yet to be established. The aim of this study is to investigate three different methods for reducing the pain and anxiety associated with the puncture of the bone marrow in adult patients. Two of the of the investigated methods involve pretreatment of the patients with pharmacological agents (sedative drug or analgetic drug), whereas the third method involves cognitive behavioural pretreatment in form of an audio material. The patients in the control group receive placebo injections.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for both first or repeated punction of the bone marrow
* Age between 18 and 85 years
* Written informed consent

Exclusion Criteria:

* Contraindication for a punction of the bone marrow
* Administration of benzodiazepines or analgetic drugs prior to the bone marrow punction
* Known hypersensitivity to benzodiazepines or Piritramid
* Known contraindication to benzodiazepines (Myasthenia gravis in particular) or Piritramid (Pheochromocytoma or conditions affecting the consciousness)
* Poor general condition (ECOG Performance Status 3,4; Karnofsky Index < 50%)
* Addictive disorders
* Administration of antidepressive drugs
* Administration of drugs that potentially depress the respiratory function
* Severe cardio-circulatory or respiratory insufficiency, sleep apnea syndrome
* Known bradycardia
* History of syncope(s) of unclear etiology
* Pregnancy or lactation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 748
Dates: Start 2001-09; Study Completion 2003-11

PRIMARY OUTCOMES:
Reduction of pain and anxiety during and after the punction procedure
Comparison of the efficacy of the three investigated methods to the placebo group, as well as to the group not receiving any pretreatment at all.

SECONDARY OUTCOMES:
Duration of the effective pain reduction in each of the investigated groups
Assessment of the quality of life in the period immediately after the bone marrow puncture

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Naumann, MD, Principal Investigator — University Clinic "Carl Gustav Carus" Dresden
Locations (1):
- Medizinische Klinik und Poliklinik I, University Clinic Carl Gustav Carus, Dresden, Saxony, Germany

REFERENCES:
- [Background] Aeschbacher BC, Portner M, Fluri M, Meier B, Luscher TF. Midazolam premedication improves tolerance of transesophageal echocardiography. Am J Cardiol. 1998 Apr 15;81(8):1022-6. doi: 10.1016/s0002-9149(98)00083-6. PMID 9576164
- [Background] Alexander JA, Smith BJ. Midazolam sedation for percutaneous liver biopsy. Dig Dis Sci. 1993 Dec;38(12):2209-11. doi: 10.1007/BF01299897. PMID 8261822
- [Background] Bein T, Tremel H, Heyde G. [Midazolam in combination with piritramid versus Thalamonal in premedication in ambulatory ENT interventions in childhood]. Anasth Intensivther Notfallmed. 1988 Aug;23(4):187-90. German. PMID 3177831
- [Background] Broome ME, Rehwaldt M, Fogg L. Relationships between cognitive behavioral techniques, temperament, observed distress, and pain reports in children and adolescents during lumbar puncture. J Pediatr Nurs. 1998 Feb;13(1):48-54. doi: 10.1016/S0882-5963(98)80068-7. PMID 9503766
- [Background] Campo R, Brullet E, Montserrat A, Calvet X, Donoso L, Bordas JM. Efficacy of low and standard midazolam doses for gastroscopy. A randomized, double-blind study. Eur J Gastroenterol Hepatol. 2000 Feb;12(2):187-90. doi: 10.1097/00042737-200012020-00009. PMID 10741933
- [Background] Chau SW, Chen CD, Yip WH, Hsu TL, Yu KL, Chang HC, Tseng CK. [Intravenous midazolam for sedation in epidural anesthesia]. Ma Zui Xue Za Zhi. 1993 Sep;31(3):157-64. Chinese. PMID 7968337
- [Background] Dahlquist LM, Power TG, Carlson L. Physician and parent behavior during invasive pediatric cancer procedures: relationships to child behavioral distress. J Pediatr Psychol. 1995 Aug;20(4):477-90. doi: 10.1093/jpepsy/20.4.477. PMID 7666289
- [Background] Dunlop TJ, Deen C, Lind S, Voyle RJ, Prichard JG. Use of combined oral narcotic and benzodiazepine for control of pain associated with bone marrow examination. South Med J. 1999 May;92(5):477-80. doi: 10.1097/00007611-199905000-00005. PMID 10342892
- [Background] Eberhart LH, Novatchkov N, Schricker T, Georgieff M, Baur CP. [Clonidine compared to midazolam for intravenous premedication for ambulatory procedures. A controlled double blind study in ASA 1 patients]. Anasthesiol Intensivmed Notfallmed Schmerzther. 2000 Jun;35(6):388-93. doi: 10.1055/s-2000-12055. German. PMID 10900497
- [Background] Ellis JA, Spanos NP. Cognitive-behavioral interventions for children's distress during bone marrow aspirations and lumbar punctures: a critical review. J Pain Symptom Manage. 1994 Feb;9(2):96-108. doi: 10.1016/0885-3924(94)90162-7. PMID 8021541
- [Background] Friedman AG, Mulhern RK, Fairclough D, Ward PM, Baker D, Mirro J, Rivera GK. Midazolam premedication for pediatric bone marrow aspiration and lumbar puncture. Med Pediatr Oncol. 1991;19(6):499-504. doi: 10.1002/mpo.2950190610. PMID 1961137
- [Background] Haberer JP. [Premedication and sedation complications during ophthalmic anesthesia]. J Fr Ophtalmol. 2000 Nov;23(9):901-6. French. PMID 11084450
- [Background] Harris CV, Bradlyn AS, Ritchey AK, Olsen BR, Pisaruk HI. Individual differences in pediatric cancer patients' reactions to invasive medical procedures: a repeated measures analysis. Pediatr Hematol Oncol. 1994 May-Jun;11(3):293-9. doi: 10.3109/08880019409141672. PMID 8060813
- [Background] Hausmann D, Wahl GH, Nadstawek J. [Analgosedation as an adjuvant during surgery under local anesthesia]. Dtsch Z Mund Kiefer Gesichtschir. 1989 Jul-Aug;13(4):246-8. German. PMID 2637069
- [Background] Jay S, Elliott CH, Fitzgibbons I, Woody P, Siegel S. A comparative study of cognitive behavior therapy versus general anesthesia for painful medical procedures in children. Pain. 1995 Jul;62(1):3-9. doi: 10.1016/0304-3959(94)00216-2. PMID 7478706
- [Background] Jay SM, Elliott CH. A stress inoculation program for parents whose children are undergoing painful medical procedures. J Consult Clin Psychol. 1990 Dec;58(6):799-804. doi: 10.1037//0022-006x.58.6.799. PMID 2292629
- [Background] Jay SM, Elliott CH, Woody PD, Siegel S. An investigation of cognitive-behavior therapy combined with oral valium for children undergoing painful medical procedures. Health Psychol. 1991;10(5):317-22. doi: 10.1037//0278-6133.10.5.317. PMID 1935866
- [Background] Kasaba T. [The effects of small dose midazolam in patients to reduce the uncomfortable feeling during epidural block procedure]. Masui. 1994 Apr;43(4):547-50. Japanese. PMID 8189620
- [Background] Korner I, Scherhag A, Preussner PR. [Analgosedation (managed anesthesia care--MAC) with propofol and piritramide for controlled cyclophotocoagulation of the eye]. Anaesthesiol Reanim. 2000;25(1):22-5. German. PMID 10721198
- [Background] Liossi C, Hatira P. Clinical hypnosis versus cognitive behavioral training for pain management with pediatric cancer patients undergoing bone marrow aspirations. Int J Clin Exp Hypn. 1999 Apr;47(2):104-16. doi: 10.1080/00207149908410025. PMID 10208073
- [Background] Mainwaring CJ, Wong C, Lush RJ, Smith JG, Singer CR. The role of midazolam-induced sedation in bone marrow aspiration/trephine biopsies. Clin Lab Haematol. 1996 Dec;18(4):285-8. PMID 9054704
- [Background] Maunuksela EL, Rajantie J, Siimes MA. Flunitrazepam-fentanyl-induced sedation and analgesia for bone marrow aspiration and needle biopsy in children. Acta Anaesthesiol Scand. 1986 Jul;30(5):409-11. doi: 10.1111/j.1399-6576.1986.tb02440.x. PMID 3766098
- [Background] Milligan DW, Howard MR, Judd A. Premedication with lorazepam before bone marrow biopsy. J Clin Pathol. 1987 Jun;40(6):696-8. doi: 10.1136/jcp.40.6.696. PMID 3611398
- [Background] Nagahama H, Okada Y, Kinouchi H, Tateda T, Aoki T, Morokawa Y. [The use of low dose midazolam for the management of spinal anesthesia]. Masui. 1997 Jun;46(6):803-8. Japanese. PMID 9223885
- [Background] Runes J, Strom C. Midazolam intravenous conscious sedation in oral surgery. A retrospective study of 372 cases. Swed Dent J. 1996;20(1-2):29-33. PMID 8738906